CLINICAL TRIAL: NCT00869427
Title: Vitamin C for Prevention of Urinary Tract Infections in the Spinal Cord Injured
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit sufficient number of patients
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sunnaas Rehabilitation Hospital, Nils Hjeltnes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 545-07286a 1.2007.2483 (REK); 2007-005657-29 (EudraCT)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-01

CONDITIONS: Urinary Tract Infection; Spinal Cord Injury
Keywords: UVI; Spinal cord injury; Prevention; Vitamin C
MeSH Terms: conditions — Urinary Tract Infections; Spinal Cord Injuries | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 vitamin C (Active Comparator): Vitamin C 1g bid
  Interventions: Drug: vitamin C
- 2 (No Intervention): Usual Care

INTERVENTIONS:
Drug: vitamin C — vitamin C 1g bid for 1 year
  Arms: 1 vitamin C

SUMMARY:
After spinal cord injury, patients have frequent urinary tract infections (UVI). Vitamin C is usually prescribed to prevent such infection, but the efficacy of the treatment is poorly documented. In the study, patients will be randomised either to receive vitamin C daily, or not, for one year, and clinical episodes of UVI will be registered. The null hypothesis is that vitamin C will not reduce the number of UVI episodes by 30%.

DETAILED DESCRIPTION:
The study is an investigator-blind randomised parallel study on the efficacy of vitamin C to prevent urinary tract infections in stable, ambulatory spinal cord-injured patients. To be included, patients should have had at least 3 previous UVI episodes over the last two years. 40 patients are included. Patients are randomised to receive either 1 g vitamin C b.i.d. over 1 year, or no vitamin C. The main outcome is the number of clinical UVIs that have been treated with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury
* 3 or more episodes of UVI over previous 2 years

Exclusion Criteria:

* pregnancy
* age <18
* continuous use of antibiotics, hippuric acid or crane berry juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Clinical episodes of UVI treated by antibiotics | one year

SECONDARY OUTCOMES:
Silent bacteriuria | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nils Hjeltnes, MD, PhD, Study Director — Sunnaas Rehabilitation Hospital